CLINICAL TRIAL: NCT01603602
Title: BOTOX® Treatment in Pediatric Upper Limb Spasticity: Double-blind Study
Brief Title: BOTOX® Treatment in Pediatric Upper Limb Spasticity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191622-101; 2012-000062-38 (EudraCT Number)
Record Dates: First submitted 2012-05-21; First posted 2012-05-22 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Pediatrics; Muscle Spasticity; Cerebral Palsy; Stroke
MeSH Terms: conditions — Muscle Spasticity; Cerebral Palsy; Stroke | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BOTOX® 3 U/kg (Experimental): Participants received intramuscular injections of BOTOX® (botulinum toxin Type A) 3 units (U) per kilogram (kg) of body weight (3 U/kg) into specified muscles of the upper limb on Day 1. Participants received weekly occupational therapy (OT).
  Interventions: Biological: botulinum toxin Type A
- BOTOX® 6 U/kg (Experimental): Participants received intramuscular injections of BOTOX® (botulinum toxin Type A) 6 U per kg of body weight (6 U/kg) into specified muscles of the upper limb on Day 1. Participants received weekly OT.
  Interventions: Biological: botulinum toxin Type A
- Placebo (Placebo Comparator): Participants received intramuscular injections of normal saline (placebo) into specified muscles of the upper limb on Day 1. Participants received weekly OT.
  Interventions: Drug: Normal Saline (Placebo)

INTERVENTIONS:
Biological: botulinum toxin Type A — Intramuscular injections of botulinum toxin Type A into specified muscles of the upper limb on Day 1.
  Other Names: BOTOX®; onabotulinumtoxinA
  Arms: BOTOX® 3 U/kg; BOTOX® 6 U/kg
Drug: Normal Saline (Placebo) — Intramuscular injections of normal saline (placebo) into specified muscles of the upper limb on Day 1.
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of BOTOX® (botulinum toxin Type A) in pediatric patients with upper limb spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Minimum weight of 10 kg/22 lb
* Upper limb spasticity due to cerebral palsy or stroke

Exclusion Criteria:

* Muscular dystrophy, myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or mitochondrial disease
* Uncontrolled epilepsy
* Botulinum Toxin therapy of any serotype for any condition within the last 6 months
* Previous surgical treatment of the study limb (except tendon lengthening), or planned surgery of the study limb during the study
* Previous casting of the study limb for spasticity within 6 months or with a dynamic splint within 3 months, or planned casting or dynamic splinting for spasticity of the study limb or affected lower limb during the study

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 235 (Actual)
Dates: Start 2012-07-12 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rozalina Dimitrova, Study Director — Allergan
Locations (45):
- United States (20):
  - AMS Neurology, Pasadena, California
  - Harrison Clinical Management, Pomona, California
  - Children's Hospital Colorado Dept. of PM&R, Aurora, Colorado
  - Associated Neurologists of Southern CT, P.C., Fairfield, Connecticut
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Axcess Medical Research, LLC, Loxahatchee Groves, Florida
  - Pediatric Neurology, PA, Orlando, Florida
  - Children's Healthcare of Atlanta Children's Rehabilitation Associates, Atlanta, Georgia
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Clinical Research Center of New Jersey, Voorhees Township, New Jersey
  - NYU Hospital for Joint Diseases, New York, New York
  - Columbia University Medical Center Dept. of Rehab. & Regenerative Medicine, New York, New York
  - OnSite Clinical Solutions, LLC, Charlotte, North Carolina
  - PMG Research if Charlotte, LLC, Charlotte, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine Texas Children's Hospital, Houston, Texas
  - Road Runner Research, San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
- Holland Bloorview Kids Rehab, Toronto, Ontario, Canada
- Debrecen University Clinical Center, Orthopedic Clinic, Debrecen, Hungary
- Philippines (2):
  - De La Salle University Medical Center, Dasmariñas, Cavite
  - Philippine Children's Medical Center, Bagong Pag-asa, Quezon City
- Poland (7):
  - Uni Centrum Kliniczne, Gdansk
  - Specjal. Gabinet Neurologiczny, Krakow
  - Centrum Medyczne "POMOC", Lodz
  - INTERMED, Lublin, Lublin
  - CRH ŻAGIEL MED, Lublin, Lublin
  - Neuro - Dzieci I Mlodziezy Aga, Warsaw
  - NZOZ Mazowieckie Centrum, Warsaw
- Russia (3):
  - Childrens Republic Hospital, Kazan'
  - Smolensk Regional Hospital- Regional Budget State Healthcare institution, Smolensk
  - Tyumen Regional Hospital #2 - State Budget Healthcare Institution of Tyumen region, Tyumen
- South Korea (6):
  - Daegu Fatima Hospital, Daegu
  - National Health Insurance Service Ilsan Hospital, Goyang-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Thailand (3):
  - Siriraj Hospital, Mahidol University, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai University, Chiang Mai
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
- Turkey (Türkiye) (2):
  - Ankara Diskapi Yildrim Beyazit, Ankara
  - Kocaeli Üniversitesi, Kocaeli

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance. — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pediatric participants with upper limb spasticity were randomized 1:1:1 to one of three treatment groups: BOTOX® 3 or 6 U/kg (unit per kilogram) or placebo.
Groups:
- BOTOX® 6 U/kg: Participants received intramuscular injections of BOTOX® (botulinum toxin Type A) 6 U/kg into specified muscles of the upper limb on Day 1. Participants received weekly occupational therapy (OT).
- BOTOX® 3 U/kg: Participants received intramuscular injections of BOTOX® (botulinum toxin Type A) 3 U/kg into specified muscles of the upper limb on Day 1. Participants received weekly OT.
Period: Overall Study
Arm/Group | BOTOX® 6 U/kg | BOTOX® 3 U/kg | Placebo
Started | 77 | 78 | 80
Completed | 75 | 78 | 79
Not Completed | 2 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Personal Reasons | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | BOTOX® 6 U/kg | BOTOX® 3 U/kg | Placebo | Total
Number analyzed (Participants) | 77 | 78 | 80 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.6 (3.66) | 8.3 (4.48) | 7.8 (4.06) | 7.9 (4.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 36 | 32 | 95
  Male | 50 | 42 | 48 | 140
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: mITT population included all randomized participants with a valid MAS-B baseline score and at least one post-baseline measurement at weeks 2, 4, or 6 for the MAS-B of the principal muscle group and the CGI by physician.
  Participants
    White: number analyzed (Participants) | 77 | 78 | 79 | 234
    White | 51 | 42 | 51 | 144
    Black: number analyzed (Participants) | 77 | 78 | 79 | 234
    Black | 3 | 3 | 3 | 9
    Asian: number analyzed (Participants) | 77 | 78 | 79 | 234
    Asian | 19 | 27 | 18 | 64
    Hispanic: number analyzed (Participants) | 77 | 78 | 79 | 234
    Hispanic | 2 | 4 | 5 | 11
    Other Unspecified: number analyzed (Participants) | 77 | 78 | 79 | 234
    Other Unspecified | 2 | 2 | 1 | 5
Modified Ashworth Scale-Bohannon (MAS-B) Score of the Principal Muscle Group Change [Mean (Standard Deviation); unit: score on a scale] — The MAS-B was used to evaluate spasticity based on grading the resistance encountered in the principal muscle group (elbow and wrist) by means of passively moving a limb through its range of motion at a study specified velocity. The resistance encountered to passive stretch was graded using a 6-point scale where: 0=no increase in muscle tone (best) to 4=affected part(s) rigid in flexion or extension (worst). For analysis purposes, the MAS-B was recoded as follows: 0=1, 1=1, 1+=2, 2=3, 3=4, 4=5. Population: Modifided Intent-to-treat (mITT) population included all randomized participants with a valid MAS-B baseline score and at least one post-baseline measurement at weeks 2, 4, or 6 for the MAS-B of the principal muscle group and the CGI by physician.
  score on a scale
    number analyzed (Participants) | 77 | 78 | 79 | 234
    (all) | 3.3 (0.45) | 3.3 (0.45) | 3.3 (0.44) | 3.3 (0.45)

OUTCOME MEASURES:

1. Primary Outcome: Average Change From Baseline in Modified Ashworth Scale-Bohannon (MAS-B) Score of the Principal Muscle Group at Weeks 4 and 6
Description: The MAS-B was used to evaluate spasticity based on grading the resistance encountered in the principal muscle group (elbow and wrist) by means of passively moving a limb through its range of motion at a study specified velocity. The resistance encountered to passive stretch was graded using a 6-point scale where: 0=no increase in muscle tone (best) to 4=affected part(s) rigid in flexion or extension (worst). For analysis purposes, the MAS-B was recoded as follows: 0=1, 1=1, 1+=2, 2=3, 3=4, 4=5. The scores at Weeks 4 and 6 were averaged. A Mixed Model Repeated Measures (MMRM) model was used for analysis. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Weeks 4 and 6
Population: Participants from the Modified Intent-to treat (mITT) population, all randomized participants with a valid MAS-B baseline score and at least one post-baseline measurement at weeks 2, 4, or 6 for the MAS-B of the principal muscle group and the CGI by physician, with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BOTOX® 6 U/kg | BOTOX® 3 U/kg | Placebo
Number analyzed (Participants) | 74 | 76 | 75
score on a scale | -1.87 (0.102) | -1.92 (0.101) | -1.21 (0.102)
Statistical Analysis 1: Comparison: BOTOX® 6 U/kg vs Placebo; Test type: Superiority; p < 0.001, Mixed Model Repeated Measures (MMRM) — MMRM model with baseline MAS-B score as covariate; factors of age, principal muscle group, treatment, visit, treatment-by-visit interaction, study center and previous botulinum toxin exposure, stratified by age and principal muscle group categories; Least Squares (LS) Mean Difference = -0.66, 95% CI 2-sided [-0.938 to -0.379]
Statistical Analysis 2: Comparison: BOTOX® 3 U/kg vs Placebo; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.71, 95% CI 2-sided [-0.992 to -0.426]

2. Primary Outcome: Average Clinical Global Impression (CGI) of Overall Change by Physician at Weeks 4 and 6
Description: The CGI of overall change (improvement or worsening) was assessed by the physician considering the participant's clinical condition and severity of side effects using a 9-point scale where: -4=very marked worsening to +4=very marked improvement. The scores at Weeks 4 and 6 were averaged. A MMRM model was used for analysis.
Time Frame: Weeks 4 and 6
Population: Participants from the m ITT population, all randomized participants with a valid MAS-B baseline score and at least one post-baseline measurement at weeks 2, 4, or 6 for the MAS-B of the principal muscle group and the CGI by physician, with data available for analysis at the given time-point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BOTOX® 6 U/kg | BOTOX® 3 U/kg | Placebo
Number analyzed (Participants) | 74 | 76 | 75
score on a scale | 1.87 (0.108) | 1.88 (0.108) | 1.66 (0.108)
Statistical Analysis 1: Comparison: BOTOX® 6 U/kg vs Placebo; Test type: Superiority; p = 0.155, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 0.21, 95% CI 2-sided [-0.082 to 0.511]
Statistical Analysis 2: Comparison: BOTOX® 3 U/kg vs Placebo; Test type: Superiority; p = 0.147, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 0.22, 95% CI 2-sided [-0.079 to 0.523]

3. Secondary Outcome: Average Change From Baseline in MAS-B Score of the Finger Flexor Muscle Group at Weeks 4 and 6
Description: The MAS-B was used to evaluate spasticity based on grading the resistance encountered in the finger flexor muscle group by means of passively moving a limb through its range of motion at a study specified velocity. The resistance encountered to passive stretch was graded using a 6-point scale where: 0=no increase in muscle tone (best) to 4=affected part(s) rigid in flexion or extension (worst). For analysis purposes, the MAS-B was recoded as follows: 0=1, 1=1, 1+=2, 2=3, 3=4, 4=5. The scores at Weeks 4 and 6 were averaged. An Analysis of Covariance (ANCOVA) model was used for analysis. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Weeks 4 and 6
Population: Participants from the mITT population, all randomized participants with a valid MAS-B baseline score and at least one post-baseline measurement at weeks 2, 4, or 6 for the MAS-B of the principal muscle group and the CGI by physician, with data available for analysis at the given time-point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BOTOX® 6 U/kg | BOTOX® 3 U/kg | Placebo
Number analyzed (Participants) | 28 | 30 | 29
score on a scale | -1.41 (0.184) | -1.46 (0.169) | -1.02 (0.170)
Statistical Analysis 1: Comparison: BOTOX® 6 U/kg vs Placebo; Test type: Superiority; p = 0.111, ANCOVA — ANCOVA model including baseline MAS-B score of finger flexor muscle group as a covariate and factors of age group, treatment group, study center, and previous botulinum toxin exposure where age group is represented by stratification categories; LS Mean Difference = -0.39, 95% CI 2-sided [-0.861 to 0.091]
Statistical Analysis 2: Comparison: BOTOX® 3 U/kg vs Placebo; Test type: Superiority; p = 0.078, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.44, 95% CI 2-sided [-0.933 to 0.051]

4. Secondary Outcome: Goal Attainment Score (GAS) as Assessed by Physician Using a 6-Point Scale
Description: Two functional goals, one active and one passive, were selected by the participant and family in consultation with the physician investigator and/or treating physical therapist relative to the lower limb impairment due to spasticity. The physician assessed the achievement of the goals using a 6-point scale: where -3=worse than start to +2=much more than expected: improvements clearly exceed the defined therapeutic goal. An ANCOVA model was used for analysis.
Time Frame: Week 8 and 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BOTOX® 6 U/kg | BOTOX® 3 U/kg | Placebo
Number analyzed (Participants) | 77 | 78 | 80
score on a scale
  Week 8, Active Goal: number analyzed (Participants) | 75 | 76 | 77
  Week 8, Active Goal | 0.11 (0.148) | 0.12 (0.148) | 0.21 (0.148)
  Week 8, Passive Goal: number analyzed (Participants) | 75 | 76 | 77
  Week 8, Passive Goal | 0.30 (0.146) | 0.23 (0.146) | 0.06 (0.146)
  Week 12, Active Goal: number analyzed (Participants) | 73 | 78 | 79
  Week 12, Active Goal | 0.49 (0.143) | 0.26 (0.139) | 0.52 (0.139)
  Week 12, Passive Goal: number analyzed (Participants) | 72 | 78 | 79
  Week 12, Passive Goal | 0.71 (0.143) | 0.31 (0.139) | 0.11 (0.139)
Statistical Analysis 1: Comparison: BOTOX® 6 U/kg vs Placebo; Week 8, Active Goal; Test type: Superiority; p = 0.636, ANCOVA — ANCOVA model including baseline MAS-B score as a covariate; factors of age, principal muscle group, treatment, study center and previous botulinum toxin exposure where age and principal muscle group were represented by stratification categories; LS Mean Difference = -0.10, 95% CI 2-sided [-0.498 to 0.305]
Statistical Analysis 2: Comparison: BOTOX® 3 U/kg vs Placebo; Week 8, Active Goal; Test type: Superiority; p = 0.658, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -0.09, 95% CI 2-sided [-0.502 to 0.318]
Statistical Analysis 3: Comparison: BOTOX® 6 U/kg vs Placebo; Week 8, Passive Goal; Test type: Superiority; p = 0.243, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 0.24, 95% CI 2-sided [-0.162 to 0.635]
Statistical Analysis 4: Comparison: BOTOX® 3 U/kg vs Placebo; Week 8, Passive Goal; Test type: Superiority; p = 0.412, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 0.17, 95% CI 2-sided [-0.237 to 0.576]
Statistical Analysis 5: Comparison: BOTOX® 6 U/kg vs Placebo; Week 12, Active Goal; Test type: Superiority; p = 0.904, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -0.02, 95% CI 2-sided [-0.408 to 0.361]
Statistical Analysis 6: Comparison: BOTOX® 3 U/kg vs Placebo; Week 12, Active Goal; Test type: Superiority; p = 0.200, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -0.25, 95% CI 2-sided [-0.641 to 0.135]
Statistical Analysis 7: Comparison: BOTOX® 6 U/kg vs Placebo; Week 12, Passive Goal; Test type: Superiority; p = 0.003, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 0.59, 95% CI 2-sided [0.210 to 0.978]
Statistical Analysis 8: Comparison: BOTOX® 3 U/kg vs Placebo; Week 12, Passive Goal; Test type: Superiority; p = 0.327, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 0.19, 95% CI 2-sided [-0.194 to 0.580]

5. Secondary Outcome: Change From Baseline in Severity of Spasticity of the Principal Muscle Group (R2-R1) Calculated Using the Modified Tardieu Scale (MTS)
Description: The MTS measured the difference between slow and fast range of motion (R2-R1) and respective change from baseline to each posttreatment office visit. The MTS of the ankle was used to determine the passive range of movement at different movement velocities, V1 (as slow as possible) and V3 (as fast as possible) with the relative difference between a slow and a fast velocity passive stretch determining the dynamic component of the muscle contracture for the joint. At each visit, the investigator measured 2 joint angles by goniometer: the R1 angle which is the angle of catch after a fast velocity (V3) stretch and the R2 angle defined as the passive joint range of movement following a slow velocity (V1) stretch. The R2 - R1 value indicated the level of the dynamic component of spasticity in the joint. The difference between slow (R2) and fast (R1) range of motion and respective change from baseline to each posttreatment office visit on the MTS was derived.
Time Frame: Baseline (Day 1) to Week 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: degrees
Arm/Group | BOTOX® 6 U/kg | BOTOX® 3 U/kg | Placebo
Number analyzed (Participants) | 77 | 78 | 80
degrees
  Change from Baseline to Week 2, Elbow: number analyzed (Participants) | 48 | 48 | 44
  Change from Baseline to Week 2, Elbow | 33.27 (5.246) | 29.58 (5.268) | 21.17 (5.602)
  Change from Baseline to Week 4, Elbow: number analyzed (Participants) | 48 | 47 | 47
  Change from Baseline to Week 4, Elbow | 31.49 (4.116) | 28.63 (4.160) | 16.78 (4.272)
  Change from Baseline to Week 6, Elbow: number analyzed (Participants) | 46 | 48 | 47
  Change from Baseline to Week 6, Elbow | 37.62 (4.372) | 28.00 (4.268) | 16.65 (4.408)
  Change from Baseline to Week 8, Elbow: number analyzed (Participants) | 47 | 48 | 48
  Change from Baseline to Week 8, Elbow | 31.17 (4.238) | 23.14 (4.188) | 15.92 (4.276)
  Change from Baseline to Week 12, Elbow: number analyzed (Participants) | 46 | 48 | 48
  Change from Baseline to Week 12, Elbow | 14.69 (3.828) | 14.06 (3.775) | 10.19 (3.854)
  Change from Baseline to Week 2, Wrist: number analyzed (Participants) | 29 | 30 | 30
  Change from Baseline to Week 2, Wrist | -15.72 (4.096) | -24.20 (3.831) | -9.60 (3.877)
  Change from Baseline to Week 4, Wrist: number analyzed (Participants) | 28 | 30 | 31
  Change from Baseline to Week 4, Wrist | -22.97 (4.965) | -25.43 (4.557) | -12.33 (4.447)
  Change from Baseline to Week 6, Wrist: number analyzed (Participants) | 28 | 30 | 30
  Change from Baseline to Week 6, Wrist | -24.33 (5.036) | -18.47 (4.641) | -7.22 (4.570)
  Change from Baseline to Week 8, Wrist: number analyzed (Participants) | 29 | 30 | 30
  Change from Baseline to Week 8, Wrist | -20.87 (4.621) | -18.90 (4.307) | -3.16 (4.303)
  Change from Baseline to Week 12, Wrist: number analyzed (Participants) | 29 | 30 | 31
  Change from Baseline to Week 12, Wrist | -16.87 (4.927) | -15.14 (4.607) | -1.62 (4.509)
Statistical Analysis 1: Comparison: BOTOX® 6 U/kg vs Placebo; Change from Baseline to Week 2, Elbow; Test type: Superiority; p = 0.117, ANCOVA — ANCOVA model including baseline MTS as a covariate and factors of age group, treatment group, study center and botulinum toxin exposure where age group is represented by stratification categories; LS Mean Difference = 12.10, 95% CI 2-sided [-3.089 to 27.293]
Statistical Analysis 2: Comparison: BOTOX® 3 U/kg vs Placebo; Change from Baseline to Week 2, Elbow; Test type: Superiority; p = 0.273, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 8.41, 95% CI 2-sided [-6.717 to 23.527]
Statistical Analysis 3: Comparison: BOTOX® 6 U/kg vs Placebo; Change from Baseline to Week 4, Elbow; Test type: Superiority; p = 0.015, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 14.71, 95% CI 2-sided [2.958 to 26.458]
Statistical Analysis 4: Comparison: BOTOX® 3 U/kg vs Placebo; Change from Baseline to Week 4, Elbow; Test type: Superiority; p = 0.046, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 11.85, 95% CI 2-sided [0.203 to 23.504]
Statistical Analysis 5: Comparison: BOTOX® 6 U/kg vs Placebo; Change from Baseline to Week 6, Elbow; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 20.97, 95% CI 2-sided [8.801 to 33.137]
Statistical Analysis 6: Comparison: BOTOX® 3 U/kg vs Placebo; Change from Baseline to Week 6, Elbow; Test type: Superiority; p = 0.064, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 11.35, 95% CI 2-sided [-0.662 to 23.362]
Statistical Analysis 7: Comparison: BOTOX® 6 U/kg vs Placebo; Change from Baseline to Week 8, Elbow; Test type: Superiority; p = 0.013, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 15.25, 95% CI 2-sided [3.317 to 27.178]
Statistical Analysis 8: Comparison: BOTOX® 3 U/kg vs Placebo; Change from Baseline to Week 8, Elbow; Test type: Superiority; p = 0.225, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 7.22, 95% CI 2-sided [-4.488 to 18.934]
Statistical Analysis 9: Comparison: BOTOX® 6 U/kg vs Placebo; Change from Baseline to Week 12, Elbow; Test type: Superiority; p = 0.409, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 4.50, 95% CI 2-sided [-6.239 to 15.236]
Statistical Analysis 10: Comparison: BOTOX® 3 U/kg vs Placebo; Change from Baseline to Week 12, Elbow; Test type: Superiority; p = 0.470, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 3.86, 95% CI 2-sided [-6.690 to 14.419]
Statistical Analysis 11: Comparison: BOTOX® 6 U/kg vs Placebo; Change from Baseline to Week 2, Wrist; Test type: Superiority; p = 0.263, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -6.13, 95% CI 2-sided [-16.962 to 4.706]
Statistical Analysis 12: Comparison: BOTOX® 3 U/kg vs Placebo; Change from Baseline to Week 2, Wrist; Test type: Superiority; p = 0.012, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -14.60, 95% CI 2-sided [-25.846 to -3.360]
Statistical Analysis 13: Comparison: BOTOX® 6 U/kg vs Placebo; Change from Baseline to Week 4, Wrist; Test type: Superiority; p = 0.098, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -10.64, 95% CI 2-sided [-23.277 to 1.996]
Statistical Analysis 14: Comparison: BOTOX® 3 U/kg vs Placebo; Change from Baseline to Week 4, Wrist; Test type: Superiority; p = 0.051, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -13.10, 95% CI 2-sided [-26.260 to 0.068]
Statistical Analysis 15: Comparison: BOTOX® 6 U/kg vs Placebo; Change from Baseline to Week 6, Wrist; Test type: Superiority; p = 0.010, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -17.11, 95% CI 2-sided [-30.031 to -4.189]
Statistical Analysis 16: Comparison: BOTOX® 3 U/kg vs Placebo; Change from Baseline to Week 6, Wrist; Test type: Superiority; p = 0.098, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -11.25, 95% CI 2-sided [-24.622 to 2.131]
Statistical Analysis 17: Comparison: BOTOX® 6 U/kg vs Placebo; Change from Baseline to Week 8, Wrist; Test type: Superiority; p = 0.005, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -17.71, 95% CI 2-sided [-29.888 to -5.537]
Statistical Analysis 18: Comparison: BOTOX® 3 U/kg vs Placebo; Change from Baseline to Week 8, Wrist; Test type: Superiority; p = 0.015, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -15.74, 95% CI 2-sided [-28.293 to -3.194]
Statistical Analysis 19: Comparison: BOTOX® 6 U/kg vs Placebo; Change from Baseline to Week 12, Wrist; Test type: Superiority; p = 0.020, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -15.25, 95% CI 2-sided [-28.010 to -2.492]
Statistical Analysis 20: Comparison: BOTOX® 3 U/kg vs Placebo; Change from Baseline to Week 12, Wrist; Test type: Superiority; p = 0.046, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -13.52, 95% CI 2-sided [-26.797 to -0.243]

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) to end of the study (Week 12)
Description: The Safety Population, all treated participants based on the treatment received, was used to determine the number of participants at risk for Serious Adverse Events and Adverse Events.
Arm/Group | BOTOX® 6 U/kg | BOTOX® 3 U/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/78 | 0/79
Serious Adverse Events (participants affected / at risk) | 3/77 | 1/78 | 1/79
Other Adverse Events (participants affected / at risk) | 15/77 | 12/78 | 17/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® 6 U/kg (N=77) | BOTOX® 3 U/kg (N=78) | Placebo (N=79)
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 0 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® 6 U/kg (N=77) | BOTOX® 3 U/kg (N=78) | Placebo (N=79)
Upper respiratory tract infection (Infections and infestations) | 7 | 4 | 2
Viral upper respiratory tract infection (Infections and infestations) | 6 | 4 | 5
Pyrexia (General disorders) | 2 | 3 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
Headache (Nervous system disorders) | 1 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT01603602/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT01603602/SAP_001.pdf